CLINICAL TRIAL: NCT03983330
Title: A Randomised Controlled Trial Evaluating the Use of Information Communication Technology (WhatsApp/WeChat) to Deliver Brief Motivational Interviewing (i-BMI) in Promoting Smoking Cessation Among Smokers With Chronic Diseases
Brief Title: Using ICT to Deliver i-BMI to Promote Smoking Cessation Among Smokers With Chronic Diseases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NTWCREC19001-2
Record Dates: First submitted 2019-05-26; First posted 2019-06-12 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The trained RA will deliver brief MI to each subject individually via WeChat or WhatsApp in the smart phones throughout the study period. The brief MI messages will be delivered more intensively as preferred by the subject (usually not less than once per 2-3 days and no more than 2 times per day) for the first 6 months. The frequency of delivering message through WeChat or WhatsApp will be interactive, depended on subjects' actions and responses.
  Start from 6 months, minimal messages by merely following the subjects' progress and responding to their questions to maintain contact will be provided to subjects till one-year follow-up.
  The readiness of quitting smoking will be assessed at 3-month follow-up. For those who are willing to take further actions to promote their health, i.e. with an intention to quit smoking, health advice on smoking will be given with more emphasis on the health benefits of quitting. The whole intervention will be given through WeChat/WhatsApp.
  Interventions: Behavioral: Brief Motivational Interviewing (i-BMI)
- Control group (Other): Subjects in the control group will not receive brief MI and follow-up booster intervention. Subjects will be informed that they will receive follow-up telephone call at 1, 3, 6 and 12 months
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Brief Motivational Interviewing (i-BMI) — The trained RA will ask the subjects about the priority of engaging in any desirable health-related lifestyle practice as identified in the completed baseline questionnaires and to state a targeted goal that they perceive as the easiest to achieve. Each subject will then receive an individual face-to-face brief MI (about 5 mins) with generic health advice on selected health-related lifestyle practice. They will then be informed to receive an individual brief MI intervention to assist behavioural changes or achieve goals as desired or chosen by them via WeChat or WhatsApp in smart phones throughout the study period. They will be given a self-help smoking cessation booklet with Hotline number.
  The RA will then deliver brief MI to each subject individually via WeChat or WhatsApp in smart phones throughout the study period.
  Readiness of quitting smoking will be assessed at 3-month follow-up. Upon request by subjects, we shall provide them with more comprehensive information on quitting.
  Arms: Intervention group
Behavioral: Control — Similar to the intervention group, the trained RA will first ask the subjects about the priority of engaging in any desirable health-related lifestyle practice and to state a targeted goal in which they perceive as the easiest to achieve after completing the baseline questionnaires. In addition, the subjects will be given a self-help smoking cessation booklet with Hotline (Tel.: 1833183). However, subjects in the control group will not receive brief MI and follow-up booster intervention. Subjects will be informed that they will receive follow-up telephone call at 1, 3, 6 and 12 months.
  Arms: Control group

SUMMARY:
To conduct a pilot study to determine the feasibility, potential efficacy and effect size of a personalized general health promotion approach using Information Communication Technology (WhatsApp or WeChat) to deliver a brief Motivational interviewing (MI) in promoting smoking cessation among smokers having follow-up in a Special Out-Patient Clinic (SOPC). In addition, this pilot study aims to assess the potential facilitators and barriers of future implementation of using such approach for smokers with chronic diseases. Based on the findings of the pilot study, a large RCT will be conducted to evaluate the effectiveness and costs of a personalized general health promotion approach in promoting smoking cessation for smokers with chronic diseases in Hong Kong in the future.

DETAILED DESCRIPTION:
Smoking has harmful effects on nearly every organ of the body and causes seven million deaths worldwide every year.1,2 Although the prevalence of daily cigarette smoking in Hong Kong has decreased from 23.3% in 1982 to 10.5 % in 2015, there are still 641,300 daily smokers3 and 400,000 hospitalisations per year that are attributable to smoking.4 Having a disease and requiring medical attention present an excellent 'teachable moment' and opportunity for initiating smoking cessation in patients, because they will be more likely to be motivated to alter their habits and improve their health. However, cigarette smoking is addictive and quitting is very difficult, with a high rate of relapse, particularly among patients with chronic diseases.5

During the past decade, we have conducted several trials on promoting smoking cessation to smokers with chronic diseases, including cardiac,6 type 2 diabetes mellitus,5 and cancer.7 We found that many smokers with chronic diseases had a long smoking history, high nicotine dependency, no quit attempt, and no intention to quit. Results of these studies indicated that about 68% smokers with cardiac diseases, 70% with diabetes mellitus and 73% with cancer recruited in Special Out-Patient Clinics (SOPC) were still in the pre-contemplation stage. We revealed that most Hong Kong smokers with chronic diseases perceived more barriers in quitting than benefits of quitting.7 Nevertheless, our previous smoking cessation interventions mostly focused on using brief interventions including stage-matched smoking cessation advices. Such interventions could be too brief and inadequate to make a great impact on such smokers. Moreover, we found that using strong warnings to communicate the risk of continued smoking might not be accepted by some of them. Hence, we need to develop and evaluate a more innovative intervention to enhance the effectiveness in promoting smoking cessation for smokers with chronic diseases. Most importantly, the new strategy should have good potential implementation in many clinical settings.

Smoking has been found to be associated with physical inactivity,8 unhealthy diet,9 and drinking.10 The interrelationship of health behaviours suggests that there could be a higher level of attribute that determines such behaviours together. Our previous studies11,12 showed that people with a general intention to promote their health are more likely to engage in desirable health-related lifestyle practices. In addition, research results showed that people once engaged in any desirable health-related lifestyle practices would progressively move to later stages of change for other health behaviours. Based on this concept, a general health promotion approach will be used to motivate smokers with intention to promote health to first engage in any desirable health-related lifestyle practices that are chosen by individual smokers, such as regular physical activity and healthy diet. It is anticipated that once they are engaged in any desirable health-related lifestyle practice they will eventually be more motivated to quit smoking.

Setting:

The study setting will be a SOPC of an acute public hospital (Tuen Mun Hospital). The Chief of Service of this unit agreed to offer support the application of this research project to be conducted in the hospital. This SOPC is chosen because of its previous participation in our RCTs on cardiac, diabetes, and cancer patients and has already been established a good collaborative relationship. In addition, Tuen Mun Hospital is one of the largest acute hospitals in Hong Kong and medical patients with chronic diseases who do not need hospitalization or are discharged will be followed up in its medical SOPC after discharging from the hospital. The capacity of this SPOC ensures the adequacy of eligible subjects to participate in this pilot study.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years or above,
* able to speak Cantonese and read Chinese
* no intention to quit smoking (pre-contemplation stage), but are willing to take action to promote health
* have a smart phone and able to use instant messaging tool (e.g. WhatsApp, WeChat) for communication, and
* willing to receive health promotion advices via WhatsApp/WeChat in the smart phone throughout the study

Exclusion Criteria:

* unable to give informed consent or participate in our intervention due to impaired mental status, cognitive impairment, or communication barrier, and
* participation in other smoking cessation programmes or services

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-11 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Biochemically validated smoking abstinence at 12 months | 12-month follow-up
  The biochemically validated 7-day point prevalence of abstinence will be confirmed by saliva cotinine level < 115 ng/ml in parallel test and a carbon monoxide level in expired air < 9 parts per million (p.p.m.).

SECONDARY OUTCOMES:
Self-reported 7-day point prevalence of smoking abstinence at 6 and 12 months | 6- and 12-month follow-up
  A structured questionnaire will be developed by adopting or modifying international and/or locally validated instruments.
Self-reported reduction of ≥ 50% in cigarette consumption at 6 and 12 months | 6- and 12-month follow-up
  A structured questionnaire will be developed by adopting or modifying international and/or locally validated instruments.
Any behavioural change reported by the subjects at 1, 3, 6 and 12 months | 1-, 3-, 6- and 12-month follow-ups
  A structured questionnaire will be developed by adopting or modifying international and/or locally validated instruments.

CONTACTS AND LOCATIONS:
Overall Officials: Ho Cheung William Li, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Li WHC, Ho LLK, Cheung AT, Wong MP, Cheung DYT, Xia W, Lam TH. A general health promotion approach to helping smokers with non-communicable diseases quit smoking: A pilot randomized controlled trial. Front Public Health. 2022 Oct 18;10:957547. doi: 10.3389/fpubh.2022.957547. eCollection 2022. PMID 36330106
- [Derived] Li WHC, Ho KY, Lam KKW, Wang MP, Cheung DYT, Ho LLK, Xia W, Lam TH. A study protocol for a randomised controlled trial evaluating the use of information communication technology (WhatsApp/WeChat) to deliver brief motivational interviewing (i-BMI) in promoting smoking cessation among smokers with chronic diseases. BMC Public Health. 2019 Aug 9;19(1):1083. doi: 10.1186/s12889-019-7417-6. PMID 31399047